CLINICAL TRIAL: NCT03388034
Title: Pertussis Immunization Programs in Low Income Countries - Ivory Coast
Acronym: PERILIC-IC
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur of Cote d'Ivoire (Other Government); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-056
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-07

CONDITIONS: Bordetella Pertussis, Whooping Cough
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal sample; Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Index case (WP1a): Infant under 6 months old with clinical signs of whooping cough syndrome.
  Nasopharyngeal sampling:
  A nasopharyngeal sample collected from each nostril by swabbing
  Interventions: Procedure: Nasopharyngeal sampling
- Control case (WP1b): Contact cases of infant with a positive diagnosis for whooping cough.
  Nasopharyngeal sampling:
  A nasopharyngeal sample collected from each nostril by swabbing
  Blood sampling:
  A blood sample collected by fingerprick
  Interventions: Procedure: Nasopharyngeal sampling; Procedure: Blood Sampling
- Seroepidemiological cohort (WP2): Children between 3 and 15 years old with complete primo-vaccination against B.Pertussis
  Blood sampling:
  A blood sample collected by fingerprick
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Nasopharyngeal sampling — A nasopharyngeal sample collected from each nostril by swabbing
  Groups: Control case (WP1b); Index case (WP1a)
Procedure: Blood Sampling — Blood sample by the tip of a finger (fingerprick)
  Groups: Control case (WP1b); Seroepidemiological cohort (WP2)

SUMMARY:
Due to waning of infectious as well as vaccine immunity and lack of vaccination boosters, a large number of adolescents and adults are no longer immunized against Bordetella pertussis, the agent of whooping cough and consequently may contract whooping cough. Furthermore, these populations represent a reservoir of the infectious agent from which the dissemination to non-immune infants is possible, causing severe illness, or even death, in this age group.

Few studies have been carried out on whooping cough in developing countries (incidence, contaminator's age, etc.) and, specifically, none have assessed the duration of protection induced by the whole cell pertussis (wP) vaccine mainly presently used in these countries.

However, data on the duration of vaccine induced protection are essential to determine i) the usefulness of vaccine boosters and ii) the target age group for these boosters.

The aims of the present study are:

* To evaluate the proportion of confirmed pertussis cases in infants presenting whooping cough syndrome (WP1a)
* To evaluate the proportion of confirmed pertussis cases or healthy carriers among contact cases
* To determine origin of the infant's contamination (WP1b)
* To determine the duration of protection induced by the wP vaccines used in contact cases and the child population aged 3 to 15 yo (WP1b and WP2)
* To bring new scientific evidences documenting the potential need for initiating boosters (WP1b and WP2)
* To allow a comparison of the results with those obtained using the same methodology for the acellular pertussis vaccine and/or in other contexts. Potential implications for the use of pertussis vaccines in low and moderate income countries.
* To increase local capabilities by the transfer of materials and expertise that will make the diagnosis of pertussis possible in the centres of reference and strengthen a pertussis monitoring network in the implicated countries.
* To improve children's health through a better match of the vaccination schedule according to the reality of the situation.

DETAILED DESCRIPTION:
Background:

Vaccination of infants and young children with a whole-cell pertussis (wP) vaccine dramatically decreased the mortality and morbidity due to B. pertussis. However, twenty-five years of "honeymoon" period, after the introduction of high vaccination coverage, reappearance of whooping cough cases in industrialized countries was observed in infants contaminated by adolescents and adults. This modification in transmission of the disease after the introduction of the wP vaccine indicated that the immunity provided by the vaccine is not lifelong, just like that provided by natural infection, and that it decreases7-9 years after the first vaccination and the first booster. Due to secondary effects, wP vaccines cannot be used for boosters. Moreover, the wP vaccines have been shown to be different in terms of efficacy (varying from 30 to 95%). Acellular pertussis (aP) vaccines consisting of purified and inactivated bacterial proteins, have therefore been developed and commercialized. These vaccines induce much fewer side effects and may therefore be used for primary-vaccination as well as for vaccine boosters. They are expensive but have more reproducible manufacturing. The humoral and long-term cell-mediated immunities granted by the aP vaccines have been shown to be comparable to the immunity granted by the wP vaccines, effective for 6-7 years after the booster vaccine in the second year of life, also inducing different cell immunity. Since 2007, the proportion of B. pertussis and B. parapertussis isolates no longer producing vaccine antigen(s) has increased in the industrialized countries that use aP vaccines. These isolates may decrease the efficacy of the aP vaccines. Does this type of isolates circulate in the Low income countries still using wP vaccines ? Does it reduce the efficacy of the wP vaccines? Moreover, the wP vaccines used in the Southern countries have not been assessed like the ones used in the Northern countries. In particular, the duration of protection after the primary-vaccination and a vaccine booster is not known.

Rational:

For various reasons, a large difference exits between the monitoring systems across the world: awareness of the disease is variable depending on the population; differences in the immunization coverage and strategies; diverse compositions of the vaccines used; but overall the large differences between the vaccines in terms of immunity against the disease, protection against infection and/or decrease in the transmission of the pathogen. The underestimation of pertussis is recognized by the World Health Organisation (WHO) and the Global Pertussis Initiative (GPI) who highlight the problem of the reliability of the declared data.

This situation is the result of i) limited use of biological diagnostics (problems in isolating the bacteria in the laboratories); ii) diagnostic errors due to the fact that diagnosis is mainly clinical ; iii) inadequate monitoring of the illness ; iv) a lack of awareness among physicians. Pertussis is not considered when it is comes to identifying the respiratory pathogen: most clinicians continue to consider it as only a child illness and ignore adult infections. The absence of an available tool allowing a reliable diagnostic to be made makes difficult to assess the real impact of this pathogen in child respiratory syndromes.

Several studies have been performed on the duration of protection induced by the wP and aP vaccines in Australia, the USA and in Europe. However, few studies have been performed on the wP vaccines used in middle and low income countries and none in Ivory Coast.

This study is part of a program entitled PERILIC which is currently conducted in Cambodia, Madagascar and Togo (NCT02983487). This research program will allow the vaccination strategy of each region concerned to be adapted when needed, as recommended by the WHO.

Expected Outcomes:

Impact on vaccination strategy:This study, as well as the analysis of data from other national programs for the surveillance of Pertussis, may raise public health authorities' awareness and help them adapting their assessment method for national vaccination programs by including the duration of protection induced by their national wP vaccine and their data on vaccine coverage, on the basis of the information in vaccination booklets, as recommended by WHO.

Impact on the improvement the children's health: The results of our study should raise the public health authorities' awareness on vaccine-preventable diseases, especially whooping cough. This raising of awareness will focus on the surveillance/monitoring and diagnosis of this disease. Moreover, the development of reliable biological diagnostic tools for pertussis will help the clinicians to confirm pertussis diagnosis and to adapt the therapeutic approach accordingly, thus improving the care of the infected person and to stop transmission of the disease which is very contagious.

Impact on the surveillance of the disease by developing an hospital-based surveillance Training, technology transfer and strengthening of the surveillance network: For the first time, the detection and identification techniques for the other species of Bordetella genus (i.e. B. parapertussis and B. holmesii) will be transferred to laboratories in Ivory Coast. The diagnosis of the different Bordetella species by real time PCR and the serological tests will be set up in the laboratories participating in this study. These laboratories could further be used by the national surveillance network and thus improve the quality of the data available for the local health authorities and for WHO. Thus, this study will allow the establishment of an effective monitoring of pertussis in Ivory Coast through the raising of the population's awareness, the training of local doctors on the clinical screening of this disease, and finally via the transfer of diagnostic techniques within the laboratories.

ELIGIBILITY:
Inclusion Criteria (Cohort 1):

* Infants under 6 months old
* Presenting clinical signs of a whooping cough syndrome
* Written consent obtained from a parent/guardian of the child

Inclusion Criteria (Cohort 2):

* People in regular and prolonged contact (>3h per day) with the index case for at least 15 days before the signs of whooping cough occurred in the infected child, living (or not) in the same household.
* For the adults, written consent obtained.
* For minors under 7 yo: written consent obtained from a parent/guardian.
* For minors over 7 yo: written consent obtained from parent/guardian and oral assent obtained from the child.

Inclusion Criteria (Cohort 3):

* Child aged between 3 and 15 yo
* Up to date first pertussis vaccination (vaccination booklet or official register)
* Last pertussis vaccination done more than one year before inclusion
* For minors under 7 yo: written consent obtained from parent/guardian.
* For minors over 7 yo: written consent obtained from parent/guardian and oral assent obtained from the child.

Exclusion Criteria (Cohort 3):

* Pertussis vaccination done more than one year before inclusion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort 1 (WP1a): Infants under 6 months old coming to hospital with clinical signs of whooping cough syndrome.
  Cohort 2 (WP1b): Contact cases of confirmed infants included in the WP1a module Cohort 3 (WP2): Children from 3 to 15 years old included, without underlying illness, with complete pertussis primo-vaccination
Sampling Method: Probability Sample
Enrollment: 789 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of biologically confirmed cases of pertussis in patients under 6 months old admitted into hospital with clinical signs corresponding to whooping cough syndrome. | December 2019
  Primary Outcome of Cohort 1 (WP1a)
Identification of the contaminator of the index case | December 2019
  Primary Outcome of Cohort 2 (WP1b)
Estimation of the protection period induced by the primo-vaccination in children between 3 and 15 yo | December 2019
  Primary Outcome of Cohort 3 (WP2)

SECONDARY OUTCOMES:
Estimation of the relative risk of the disease occurring in the contact patients based on their immunization status and age groups | June 2020

CONTACTS AND LOCATIONS:
Overall Officials: Fabien TAIEB, MD, MSc, MPH, Principal Investigator — Institut Pasteur; Man-Koumba SOUMAHORO, PhD, Principal Investigator — Institut Pasteur of Cote d'Ivoire; Nicole GUISO, PhD, Study Chair — Institut Pasteur
Locations (5):
- Côte d’Ivoire (5):
  - Centre de Santé Urbain à base Communautaire (CSU-Com) d'Angré, Abidjan
  - CHU d'Angré, Abidjan
  - Hôpital Général de Port-Bouët, Abidjan
  - Hôpital Général de Yopougon Attié, Abidjan
  - Institut Pasteur de Côte d'Ivoire, Abidjan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guiso N, Wirsing von Konig CH. Surveillance of pertussis: methods and implementation. Expert Rev Anti Infect Ther. 2016 Jul;14(7):657-67. doi: 10.1080/14787210.2016.1190272. Epub 2016 May 31. PMID 27224518
- [Background] Tubiana S, Belchior E, Guillot S, Guiso N, Levy-Bruhl D; Renacoq Participants. Monitoring the Impact of Vaccination on Pertussis in Infants Using an Active Hospital-based Pediatric Surveillance Network: Results from 17 Years' Experience, 1996-2012, France. Pediatr Infect Dis J. 2015 Aug;34(8):814-20. doi: 10.1097/INF.0000000000000739. PMID 25955837
- [Background] Guiso N. Pertussis vaccination and whooping cough: and now what? Expert Rev Vaccines. 2014 Oct;13(10):1163-5. doi: 10.1586/14760584.2014.941816. Epub 2014 Jul 14. PMID 25020131
- [Background] Heininger U, Andre P, Chlibek R, Kristufkova Z, Kutsar K, Mangarov A, Meszner Z, Nitsch-Osuch A, Petrovic V, Prymula R, Usonis V, Zavadska D. Comparative Epidemiologic Characteristics of Pertussis in 10 Central and Eastern European Countries, 2000-2013. PLoS One. 2016 Jun 3;11(6):e0155949. doi: 10.1371/journal.pone.0155949. eCollection 2016. PMID 27257822
- [Background] Guiso N, Levy C, Romain O, Guillot S, Werner A, Rondeau MC, Bechet S, Cohen R. Whooping cough surveillance in France in pediatric private practice in 2006-2015. Vaccine. 2017 Oct 27;35(45):6083-6088. doi: 10.1016/j.vaccine.2017.09.072. Epub 2017 Sep 30. PMID 28974408
- [Background] von Koenig CHW, Guiso N. Global burden of pertussis: signs of hope but need for accurate data. Lancet Infect Dis. 2017 Sep;17(9):889-890. doi: 10.1016/S1473-3099(17)30357-2. Epub 2017 Jun 13. No abstract available. PMID 28623145